CLINICAL TRIAL: NCT06475183
Title: Effects of Probiotics on Inflammatory Biomarkers in Persons With Multiple Sclerosis (MS) and in Family Members of Persons With MS
Brief Title: Probiotic Chocolate Study in Multiple Sclerosis
Acronym: ProChocolate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAU8857
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Healthy Nutrition
Keywords: muliple sclerosis; probiotic
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probioitic consumption (Experimental): All pariticpants will consume Bouchard Belgian Dark Chocolate Probiotic Napolitains, containing bifidobacterium longum in a quantity of 10 billium CFUs daily
  Interventions: Dietary Supplement: Bouchard Belgian Dark Chocolate Probiotic Napolitains, containing bifidobacterium longum

INTERVENTIONS:
Dietary Supplement: Bouchard Belgian Dark Chocolate Probiotic Napolitains, containing bifidobacterium longum — Bouchard Belgian Dark Chocolate Probiotic Napolitains containing 10 billion CFUs of bifidobacterium longum daily for 6 weeks

SUMMARY:
The goal of this study is to assess the effects of probiotics on persons with multiple sclerosis (MS), persons at higher genetic risk for MS (first degree family members of persons with MS), and healthy controls. Participants will be asked to consume probiotic containing chocolates (Bouchard Belgian Dark Chocolate Probiotic Napolitains containing 10 billion CFUs of bifidobacterium longum per day) for 6 weeks. Participants will undergo blood draws before and after the 6 weeks of probiotic containing chocolate and microbial metabolites and immune markers will be compared before and after the probiotics, as well as between groups.

DETAILED DESCRIPTION:
The goal of this study is to assess the effects of probiotics in persons with MS (PwMS), persons at high genetic risk for MS (first degree family members of PwMS), and healthy controls. PwMS. Subjects undergo blood draws and will complete surveys on neurological symptoms (as relevant). Subjects are given a supply of individually wrapped probiotic containing chocolates (Bouchard Belgian Dark Chocolate Probiotic Napolitains) along with instructions on proper storage, dosage, and a diary to complete regarding supplement adherence. After a "ramp up" period of 3 days during which participants will consume take 2 chocolates per day, participants consume 5 chocolates per day (10 billion CFUs of bifidobacterium longum per day) for 6 weeks. After 6 weeks participants return the adherence diaries and answer questions about probiotic tolerance. They also repeat similar surveys and again undergo blood draws. Serum levels of microbial metabolites and peripheral blood immune profiles are assessed before and after supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis (MS) subjects, first-degree relatives of MS subjects, or healthy controls
* Age 18-45

Exclusion Criteria:

* diabetes
* tree nut allergy
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
peripheral blood mononuclear cell (PBMC) profile: Change in Regulatory T (Treg) cells | baseline (week 0) to week 6
  percent change in Treg cells from baseline to week 6
peripheral blood mononuclear cell (PBMC) profile: Change in T helper (TH) cells | baseline (week 0) to week 6
  change in ratio of TH1 to Th2 cells from baseline to week 6
peripheral blood mononuclear cell (PBMC) profile: Change in T helper Th17 cells | baseline (week 0) to week 6
  percent change in Th17 cells from baseline to week 6
Change in serum microbial metabolites | baseilne (week 0) to week 6
  percent change in short chain fatty acid levels from baseline to week 6

SECONDARY OUTCOMES:
Change in Modified Fatigue Impact Scale-5 Impact Scale | week 0, week 6
  brief patient reported measure of fatigue, range of values is 0-20 with a higher score indicating worse outcome
Change in Patient-Determined Disability Scale (PDDS) | week 0, week 6
  brief-patient reported meausre of disability in MS, range of values is 0-8 with higher score indicating worse outcome
Change in Bowel Control Scale | week 0, week 6
  brief patient reported measure of bowel control and impact of bowel problems on everyday life, range of scores is 0-16 with higher score indicating worse outcome
Change in Multiple Sclerosis Rating Scale- Revised (MSRS-R) Patient-Determined Disease Steps Scale | week 0, week 6
  brief patient reported measure of disability in MS, range of scores is 0-32 with higher score indicating higher disability

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Straus Farber, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No